CLINICAL TRIAL: NCT04503902
Title: A Multi-center, Open, Dose Exploration and Dose Expansion Phase I/II Clinical Study of Toripalimab（JS001） Combined With Donafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Toripalimab Combined With Donafenib in the Treatment of Advanced Hepatocellular Carcinoma
Acronym: HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001D-C-102
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: interventions — donafenib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001+Donafenib (Experimental): Donafenib 100mg QD/100 mg BID/200 mg BID orally + JS001 240mg Q3W iv
  Interventions: Drug: Donafenib Tosilate Tablets; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: Donafenib Tosilate Tablets — In the dose exploration phase (phase I)，three doses of Donafenib tosylate tablets [100 mg once a day (QD); 100 mg twice a day (BID); 200 mg, BID] will be explored. In the dose expansion phase (phase II), patients will be treated at the recommended dose for phase 2(RP2D).The RP2D will be determined by the dose escalation study.
  Other Names: Donafenib
Drug: Toripalimab Injection — JS001 will be administrated by intravenous (i.v.) infusion once every 21 days
  Other Names: JS001

SUMMARY:
This study is an open, multi-center phase I/II clinical study.

DETAILED DESCRIPTION:
It will explore the tolerability (phase I) and effectiveness (phase II) of the Donafenib tosilate tablets combined with Toripalimab injection in patients with advanced HCC. The study is conducted in two phases, the first phase is the dose exploration phase (phase I), and the second phase is the dose expansion phase (phase II).

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic HCC who are not suitable for surgical resection, who are clinically diagnosed or confirmed by histopathology and/or cytology according to the "Standards for the Diagnosis and Treatment of Primary Liver Cancer" (2017);
* At least one measurable lesion (according to RECIST v1.1);
* ECOG performance status score of 0 or 1;
* Life expectancy ≥ 12 weeks；
* Have not received systemic therapy (systemic chemotherapy and/or molecular targeted therapy).If the patient has received adjuvant chemotherapy after local treatment, the chemotherapy needs to be over for more than 12 months, and disease progression or metastasis occurs；
* Fully understand this research and voluntarily sign the ICF。

Exclusion Criteria:

* Patients with diffuse liver cancer, hepatic encephalopathy that is difficult to control, and liver cancer patients whose lesion size accounts for 70% or more of the entire liver.
* Patients with intrahepatic cholangiocarcinoma (ICC) or HCC-ICC mixed type；
* Tumor invades inferior vena cava VP4.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after the first dose of JS001 and Donafenib
  Severe toxicity that may be related to JS001 or donafenib during dose escalation of phase I clinical trial
Objective response rate（ORR） as determined by the Invertigator using RECIST V1.1 | From the time of initial administration until intolerant toxicity, disease progression, withdrawal of ICF, loss of follow-up, death or early study termination occurs (whichever occurs first),assessed up to 18 months
  The ratio of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Anti-JS001 antibody | From the time of initial administration until intolerant toxicity, disease progression, withdrawal of ICF, loss of follow-up, death or early study termination occurs (whichever occurs first),assessed up to 18 months
Overall survival (OS) | From the time of initial administration until intolerant toxicity, disease progression, withdrawal of ICF, loss of follow-up, death or early study termination occurs (whichever occurs first),assessed up to 18 months
  The Kaplan-Meier survival from the initiation date of first cycle until death from any cause or the last follow-up date.
Progression free survival (PFS) | From the time of initial administration until intolerant toxicity, disease progression, withdrawal of ICF, loss of follow-up, death or early study termination occurs (whichever occurs first),assessed up to 18 months
  The Kaplan-Meier survival from the initiation date of first cycle until the date of first documented progression or date of death

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, PhD, Principal Investigator — No.81 Hospital of PLA
Locations (1):
- No.81 Hospital of PLA, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No